CLINICAL TRIAL: NCT04005053
Title: Identifying Biological Signatures of N-Acetylcysteine for Non-Suicidal Self-Injury in Adolescents and Young Adults
Brief Title: Signatures of N-Ac for Non-Suicidal Self-Injury in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26890
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Self-Harm; Depression; Suicide
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Suicide | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-Dose NAC (Experimental): 3600 NAC mg/day
  Interventions: Drug: N-acetyl cysteine
- High-Dose NAC (Experimental): 5400 NAC mg/day
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: N-acetyl cysteine — 3600 or 5400 mg/day N-acetyl cysteine
  Other Names: N-acetylcysteine
  Arms: High-Dose NAC; Low-Dose NAC
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
To measure NAC-induced changes to concentrations of glutathione (GSH) in the anterior cingulate cortex (ACC) as measured by magnetic resonance spectroscopy (MRS) in 36 adolescents and young adults with NSSI (12 in each group: high, low, and placebo).

DETAILED DESCRIPTION:
This study is a double-blind, placebo controlled, 4-week course of two-tiered N-acetylcysteine (NAC) dosing focused on identifying the optimal dose to achieve meaningful change in measurable biomarkers (glutathione and glutamate).

This design will allow us to confirm acute biological changes, select the optimal dose for achieving biological effects, and examine dose/concentration-response relationships with respect to biological markers and pharmacokinetics.

Brief schedule of activities: Subjects will be recruited through community and clinical settings and screened over the phone. There will be a total of 4 in-person visits and two sets of on-line study activities.

Eligible participants will be assigned to one of 3 groups (double-blinded): a low-dose NAC group (3600 mg/day), a high-dose NAC group (5400mg/day), and placebo (PBO). The study intervention period is 4 weeks. Total participation is up to 8 weeks, depending on the length of time between Day 0 and Day 1.

The investigators will recruit 36 adolescents and young adults aged 16-24 years. There will be 12 participants in each group (PBO, 3600mg/day, 5400mg/day). The investigators will use a minimization procedure to ensure that the participants in these 3 groups will have similar age, clinical severity and medication status.

ELIGIBILITY:
Inclusion Criteria:

* Current frequency of at least one NSSI episode in the past 2 months
* ≥ 5 past episodes of NSSI with significant tissue damage (e.g. scars present)
* Psychotropic medications are dose-stable for 1 month
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Any MRI contraindications (e.g. metal plates, claustrophobia, braces, implanted devices)
* Any current serious medical illness as defined by medical history
* Current Substance Use Disorder (except Tobacco Use Disorder)
* Primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, schizophreniform disorder)
* Neurodevelopmental disorder such as mental retardation or autism
* Changes in psychotropic medications in past 1 month
* Taken NAC or glutathione on a regular basis in the past 6 months
* Currently pregnant, planning to become pregnant, currently breastfeeding, or unwillingness to use contraception throughout the study.
* Allergy/sensitivity to N-acetylcysteine.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahasrabudhe SA, Silamongkol T, Park YW, Colette A, Eberly LE, Klimes-Dougan B, Coles LD, Cloyd JC, Oz G, Mueller BA, Kartha RV, Cullen KR. Identifying Biological Signatures of N-Acetylcysteine for Non-Suicidal Self-Injury in Adolescents and Young Adults. J Psychiatr Brain Sci. 2021;6:e210007. doi: 10.20900/jpbs.20210007. Epub 2021 Apr 29. PMID 34036177

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo
Started | 16 | 13 | 15
Completed | 14 | 11 | 14
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo | Total
Number analyzed (Participants) | 14 | 11 | 14 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2) | 21 (2) | 21 (2) | 21 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 14 | 39
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 9 | 11 | 30
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Increase in Glutathione (GSH) Concentrations in the ACC
Description: increase in glutathione (GSH) concentrations in the anterior cingulate cortex (ACC) as measured by magnetic resonance spectroscopy (MRS)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo
Number analyzed (Participants) | 14 | 11 | 14
Percent change | 5 (12) | 0 (10) | 2 (15)

2. Secondary Outcome: Change in GSH Reduced-to-oxidized Ratio
Description: Percent increase in reduced-to-oxidized ratio of glutathione (GSH) in the blood compared to baseline
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo
Number analyzed (Participants) | 14 | 11 | 14
percent change | 14 (15) | 28 (51) | -5 (26)

3. Secondary Outcome: Change in Glutamate Concentrations
Description: Percent decrease in the concentrations of glutamate (GLU) in the anterior cingulate cortex (ACC) measured by MRS
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo
Number analyzed (Participants) | 14 | 11 | 14
percent change | -0.9 (2.6) | -1.2 (4.2) | -0.8 (4.6)

ADVERSE EVENTS:
Time Frame: recorded by study staff throughout the study occurring any time after informed consent is obtained for 8 weeks.
Arm/Group | Low-Dose NAC | High-Dose NAC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11 | 1/14
Other Adverse Events (participants affected / at risk) | 10/14 | 9/11 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose NAC (N=14) | High-Dose NAC (N=11) | Placebo (N=14)
Hospitalization due to suicidality (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose NAC (N=14) | High-Dose NAC (N=11) | Placebo (N=14)
Psychiatric (Psychiatric disorders) | 5 (7) | 4 (5) | 5 (8)
Gastrointestinal (Gastrointestinal disorders) | 5 (5) | 5 (6) | 3 (4)
Cardiovascular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Nervous system (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
ENT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04005053/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04005053/ICF_001.pdf